CLINICAL TRIAL: NCT02613741
Title: Metabolism of Fibrinogen and Apolipoprotein B-100 in Childhood Obesity and Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Babu Balagopal, Director, Biomedical Analysis Laboratory, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C.20.8840; 0030342B (Other Grant/Funding Number: American AHeart Association)
Record Dates: First submitted 2015-11-19; First posted 2015-11-24 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Obesity; Cardiovascular Disease
MeSH Terms: conditions — Obesity; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): 12 weeks of lifestyle-based physical activity intervention
  Interventions: Other: Lifestyle-based physical activity
- Control (No Intervention): 12 weeks of no intervention

INTERVENTIONS:
Other: Lifestyle-based physical activity — Obese subjects will undergo a randomized physical activity-based weight reduction program (12 weeks). The lifestyle intervention will be determined based on an initial evaluation of each subjects' energy expenditure (by indirect calorimetry). Caloric intake will be set to elicit the loss of 1 to 1.5 lbs/week. The subjects and the family will meet with a dietitian once/week for 12 weeks. The intervention group will undergo an aerobic exercise program 3 times/week. The duration of exercise will be progressively increased from 20 to 45 minutes/session. The subjects will keep daily record of exercise activity and food intake. Interventions will be monitored during the subjects' weekly visit with the research group and they will be given counseling to stick to the intervention program.
  Arms: Intervention

SUMMARY:
Since obesity and plasma fibrinogen levels are important CVD risk factors in the adults, and since childhood obesity is a major risk factor for adult obesity and also because it is not established whether or not this is due to an increase in the FSR of fibrinogen, the investigators set up the studies with the following specific aims:

1. To investigate the metabolism of fibrinogen and VLDL apoB-100, CVD risk factors, in childhood obesity by measuring their fractional synthetic rate (FSR) compared to lean age and sex matched controls
2. To determine the outcome of a three month non-pharmacological intervention (physical exercise combined with controlled diet) to reduce weight on the FSR of fibrinogen and apoB-100
3. To determine the relationship between FSR of fibrinogen and IL-6 in obese children and its potential implications on CVD before and after the non-pharmacological intervention
4. To determine other CVD risk factors, PAI-1 levels, D-Dimer concentration, homocysteine, insulin, free fatty acid, HDL & LDL cholesterol and blood pressure in response to weight reduction (as consequence of a combined program of diet and exercise).

DETAILED DESCRIPTION:
A. SPECIFIC AIMS:

Evidence from the literature suggests that:

1. childhood onset of obesity increases the risk of obesity and cardiovascular disease (CVD) in adulthood;
2. plasma fibrinogen and apolipoprotein B-100 (apoB-100) levels are elevated in obesity;
3. elevated levels of plasma fibrinogen and apolipoprotein B-100 (apoB-100) are major independent risk factors for CVD in adults;
4. raised plasma fibrinogen levels in obese children and/adolescents could be a major factor responsible for CVD morbidity and mortality in adulthood;
5. a low level of physical activity is associated with a high level of plasma fibrinogen in adults;
6. physical training and controlled diet have been proved to be non-pharmacological ways to improve hemostatic function in adults, thereby reducing heart disease risk. Despite these evidences the mechanism of these changes remain unclear. A better understanding of the mechanism of these changes will lead to more directed therapies to reduce these risk factors early in life.

The increased plasma concentrations of fibrinogen (and/or other proteins) is decided by the equilibrium between two dynamic processes in the body, namely, synthesis and degradation rates of these proteins. Therefore, elevated levels of fibrinogen must be a consequence of:

1. increased fibrinogen synthesis;
2. decreased fibrinogen degradation or
3. a contribution of both.

For designing effective therapies it is important to know, whether the increased concentration of plasma fibrinogen is due to increased synthesis or decreased degradation or both. Using stable isotope mass spectrometry techniques it is possible to measure the synthesis rates of proteins in vivo in humans. Yet until now there are no reports on the direct measurement of FSR of fibrinogen and/or apoB-100 in childhood obesity, important CVD risk factors. The direct measurement of degradation rates of proteins in vivo in humans, however, is not easily done. Few studies have reported changes in the concentrations of fibrinolytic markers such as plasminogen activator inhibitor-1 (PAI-1) and D-Dimer in obesity. This, however, accounts for only a small fraction of the elevated levels of plasma fibrinogen in childhood obesity. On the other hand recent preliminary results in three subjects from our lab show that fibrinogen synthesis rate is substantially higher (more than two times) in obese adolescent girls Vs lean controls (please see results under "Preliminary results" below). Pro-inflammatory cytokines, particularly interleukin-6 (IL-6), are known to play an important role in the regulation of acute phase reactive proteins associated with inflammation, including fibrinogen. A direct link between IL-6 and increased FSR of plasma fibrinogen in childhood obesity and CVD, however, is unknown. Also, other mechanisms involving insulin resistance and free fatty acid/albumin ratio are also equally plausible for the increased synthesis of fibrinogen in obesity and CVD. Therefore, it is important to understand and establish the relationship between increased FSR of fibrinogen and these regulating factors in this study for two reasons:

1. to better design effective therapies based on these results and
2. to further understand the pathophysiology of these changes in CVD and obesity.

The overall purpose of the proposed studies is therefore:

1. to expand on our preliminary data and establish the observation of increased fibrinogen synthesis rate (in three subjects) in childhood obesity
2. to understand the relationship between increased FSR of fibrinogen and changes IL-6, insulin and glucose levels and free fatty acid (FFA) levels and FFA/albumin ratio in obese vs lean children
3. to study the effect of a non-pharmacological intervention program for three months (12 weeks), that involves weight reduction due to exercise and controlled diet on fibrinogen, apoB-100 and other cardiovascular risk factors and their relationship to changes in IL-6 levels, insulin/glucose ratio (a measure of insulin resistance), FFA/albumin ratio.

The proposed grant will use in vivo stable isotope (non-radioactive) dilution techniques, to test the following hypothesis:

Hypotheses:

1. higher rates of synthesis of fibrinogen and apoB-100 contribute substantially to their elevated levels in obese children;
2. plasma fibrinogen and apoB-100 concentration and synthesis decrease by non-pharmacological intervention to reduce weight, that involves regular physical exercise and controlled diet;
3. IL-6 and/or insulin resistance are important mechanistic links between increased plasma fibrinogen FSR and increased CVD risk and obesity and
4. the non-pharmacological intervention program modulates other CVD risk factors such as PAI-1, D-Dimer, homocysteine, free fatty acids, insulin, glucose, HDL and LDL cholesterol levels and IL-6 concentrations along with fibrinogen synthesis.

Summary of Specific Aims

Since obesity and plasma fibrinogen levels are important CVD risk factors in the adults, and since childhood obesity is a major risk factor for adult obesity and also because it is not established whether or not this is due to an increase in the FSR of fibrinogen, the investigators set up the studies with the following specific aims:

1. To investigate the metabolism of fibrinogen and VLDL apoB-100, CVD risk factors, in childhood obesity by measuring their fractional synthetic rate (FSR) compared to lean age and sex matched controls
2. To determine the outcome of a three month non-pharmacological intervention (physical exercise combined with controlled diet) to reduce weight on the FSR of fibrinogen and apoB-100
3. To determine the relationship between FSR of fibrinogen and IL-6 in obese children and its potential implications on CVD before and after the non-pharmacological intervention
4. To determine other CVD risk factors, PAI-1 levels, D-Dimer concentration, homocysteine, insulin, free fatty acid, HDL & LDL cholesterol and blood pressure in response to weight reduction (as consequence of a combined program of diet and exercise).

ELIGIBILITY:
Inclusion Criteria:

* Obese: BMI ≥30 kg/m2
* Lean (controls): BMI ≤ 25 kg/m2) age 14 to 18 years and Tanner stage matched
* Ability to understand and cooperate with the procedures
* Signed informed consent from subjects and parents

Exclusion Criteria:

* Medications such as Beta-adrenergic blockers, steroids and other drugs known to affect protein metabolism
* Heart disease
* Chronic liver disease
* Chronic renal disease
* Active malignancy
* Alcoholism or drug abuse
* Anemia
* Inter-current illness over the 7 days before the study
* Surgery in the past 3 months

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2001-01 (Actual); Primary Completion 2004-01 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Protein turnover | 12 weeks
  Stable isotope mass spectrometry
Fractional synthesis rate of fibrinogen | 12 weeks
  Stable isotope mass spectrometry
Fibrinogen | 12 weeks
  Plasma concentration measured by nephelometry

SECONDARY OUTCOMES:
Fat mass | 12 weeks
  Dual-energy X-ray absorptiometry (DEXA)
Fat free mass | 12 weeks
  Dual-energy X-ray absorptiometry (DEXA)

CONTACTS AND LOCATIONS:
Overall Officials: Babu Balagopal, PhD, Principal Investigator — Nemours Children's Clinic

REFERENCES:
- [Result] Balagopal P, Bayne E, Sager B, Russell L, Patton N, George D. Effect of lifestyle changes on whole-body protein turnover in obese adolescents. Int J Obes Relat Metab Disord. 2003 Oct;27(10):1250-7. doi: 10.1038/sj.ijo.0802388. PMID 14513074
- [Result] Balagopal P, George D, Patton N, Yarandi H, Roberts WL, Bayne E, Gidding S. Lifestyle-only intervention attenuates the inflammatory state associated with obesity: a randomized controlled study in adolescents. J Pediatr. 2005 Mar;146(3):342-8. doi: 10.1016/j.jpeds.2004.11.033. PMID 15756217
- [Result] Balagopal P, George D, Yarandi H, Funanage V, Bayne E. Reversal of obesity-related hypoadiponectinemia by lifestyle intervention: a controlled, randomized study in obese adolescents. J Clin Endocrinol Metab. 2005 Nov;90(11):6192-7. doi: 10.1210/jc.2004-2427. Epub 2005 Aug 30. PMID 16131584
- [Result] Balagopal P, Graham TE, Kahn BB, Altomare A, Funanage V, George D. Reduction of elevated serum retinol binding protein in obese children by lifestyle intervention: association with subclinical inflammation. J Clin Endocrinol Metab. 2007 May;92(5):1971-4. doi: 10.1210/jc.2006-2712. Epub 2007 Mar 6. PMID 17341558
- [Result] Balagopal P, George D, Sweeten S, Mann KJ, Yarandi H, Mauras N, Vaughan DE. Response of fractional synthesis rate (FSR) of fibrinogen, concentration of D-dimer and fibrinolytic balance to physical activity-based intervention in obese children. J Thromb Haemost. 2008 Aug;6(8):1296-303. doi: 10.1111/j.1538-7836.2008.03037.x. Epub 2008 May 26. PMID 18507721
- [Result] Balagopal PB, Gidding SS, Buckloh LM, Yarandi HN, Sylvester JE, George DE, Funanage VL. Changes in circulating satiety hormones in obese children: a randomized controlled physical activity-based intervention study. Obesity (Silver Spring). 2010 Sep;18(9):1747-53. doi: 10.1038/oby.2009.498. Epub 2010 Jan 21. PMID 20094040
- [Result] Lovely R, Hossain J, Ramsey JP, Komakula V, George D, Farrell DH, Balagopal PB. Obesity-related increased gamma' fibrinogen concentration in children and its reduction by a physical activity-based lifestyle intervention: a randomized controlled study. J Pediatr. 2013 Aug;163(2):333-8. doi: 10.1016/j.jpeds.2013.01.004. Epub 2013 Feb 14. PMID 23415619
- [Derived] Cosentino RG, Churilla JR, Josephson S, Molle-Rios Z, Hossain MJ, Prado WL, Balagopal PB. Branched-chain Amino Acids and Relationship With Inflammation in Youth With Obesity: A Randomized Controlled Intervention Study. J Clin Endocrinol Metab. 2021 Oct 21;106(11):3129-3139. doi: 10.1210/clinem/dgab538. PMID 34286837